CLINICAL TRIAL: NCT06587451
Title: A Randomized, Double-blind, Parallel-group Study to Compare Pharmacokinetics, Efficacy, Safety, and Immunogenicity of JPB898 (Proposed Nivolumab Biosimilar) and US-licensed and EU-authorized Opdivo® in Combination With Yervoy® in Participants With Untreated Advanced (Unresectable/Metastatic) Melanoma
Brief Title: Integrated Pharmacokinetics (PK)/Efficacy, Safety, and Immunogenicity Study to Demonstrate Similarity of JPB898, a Proposed Biosimilar to Nivolumab, to Opdivo® in Combination With Yervoy®
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: In light of the evolving regulatory landscape and growing indications that major Health Authorities will move towards a streamlined clinical development, Sandoz took a strategic decision and is winding down its CJPB898A12301 clinical study.
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CJPB898A12301
Record Dates: First submitted 2024-08-30; First posted 2024-09-19 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Neoadjuvant Therapy; Maintenance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- JPB898 (Experimental): Participants will receive JPB898 combined with Yervoy-EU during the induction phase. Participants will receive JPB898 during maintenance phase.
  Interventions: Drug: JPB898 (Induction and Maintenance); Drug: Yervoy-EU (Induction)
- Opdivo-EU (Active Comparator): Participants will receive Opdivo-EU combined with Yervoy-EU during the induction phase. Participants will receive Opdivo-EU during the maintenance phase.
  Interventions: Drug: Opdivo-EU (Induction); Drug: Yervoy-EU (Induction); Drug: Opdivo-EU (Maintenance)
- Opdivo-US (Active Comparator): Participants will receive Opdivo-US combined with Yervoy-EU during the induction phase. Participants will receive Opdivo-EU during the maintenance phase.
  Interventions: Drug: Opdivo-US (Induction); Drug: Yervoy-EU (Induction); Drug: Opdivo-EU (Maintenance)

INTERVENTIONS:
Drug: JPB898 (Induction and Maintenance) — Induction and Maintenance: Intravenous (IV)
  Arms: JPB898
Drug: Opdivo-EU (Induction) — Induction: Intravenous (IV)
  Arms: Opdivo-EU
Drug: Opdivo-US (Induction) — Induction: Intravenous (IV)
  Arms: Opdivo-US
Drug: Yervoy-EU (Induction) — Induction: Intravenous (IV)
Drug: Opdivo-EU (Maintenance) — Maintenance: Intravenous (IV)
  Arms: Opdivo-EU; Opdivo-US

SUMMARY:
The purpose of the study is to demonstrate similar PK and efficacy and to show comparable safety and immunogenicity between JPB898, Opdivo-EU, and Opdivo-US, all administered in combination with Yervoy-EU (induction phase only), in participants with advanced (unresectable Stage III or metastatic Stage IV) melanoma.

ELIGIBILITY:
Inclusion Criteria

* Male or female participants must be 18 years or older.
* Histologically confirmed melanoma.
* Unresectable or metastatic melanoma measurable by Computerized tomography (CT) or Magnetic resonance imaging (MRI).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Known Programmed cell death ligand 1 (PD-L1) and BRAF mutational status or consent to testing.
* Sexually active participants must agree to use effective contraception.

Exclusion Criteria

* Active brain or leptomeningeal metastases unless stable for 8 weeks.
* Ocular melanoma.
* Prior active malignancy within the last year untreated or still requiring treatment.
* Severe and uncontrolled conditions, active Hepatitis B/C, Human immunodeficiency virus (HIV), or autoimmune diseases requiring systemic treatment.
* Previous treatment with specific immune checkpoint inhibitors, systemic anticancer therapy, or radiotherapy for melanoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Demonstrate PK similarity between JPB898, Opdivo-US, and Opdivo-EU | Days 1 to 22
  Area under the serum concentration-time curve measured from the time of dosing of the first dose to the second dose (AUCtrunc) after the first dose
Demonstrate PK similarity between JPB898, Opdivo-US, and Opdivo-EU between JPB898 and Opdivo-US/-EU | Days 64 to 85
  Area under the serum concentration-time curve measured from the time of dosing to the last measurable serum concentration in the dosing interval, tau (AUCtau) after the fourth dose
Demonstrate efficacy similarity for Best overall response (BOR) between JPB898 and Opdivo-US/-EU defined as the best overall response based on blinded central tumor assessments using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria | BOR (Complete response (CR) or partial response (PR)) from baseline up to 28 weeks
  The assessment of response for the primary efficacy is based on tumor response data as per blinded independent central review and according to RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (57):
- Sandoz Investigational Site, Sofia, Bulgaria
- Chile (3):
  - Sandoz Investigational Site, Providencia
  - Sandoz Investigational Site, Santiago
  - Sandoz Investigational Site, Viña del Mar
- Georgia (2):
  - Sandoz Investigational Site, Batumi
  - Sandoz Investigational Site, Tbilisi
- Germany (3):
  - Sandoz Investigational Site, Chemnitz
  - Sandoz Investigational Site, Düsseldorf
  - Sandoz Investigational Site, Giessen
- Greece (2):
  - Sandoz Investigational Site, Athens
  - Sandoz Investigational Site, Thessaloniki
- Italy (8):
  - Sandoz Investigational Site, Bari
  - Sandoz Investigational Site, Meldola
  - Sandoz Investigational Site, Pisa
  - Sandoz Investigational Site, Ravenna
  - Sandoz Investigational Site, Roma
  - Sandoz Investigational Site, Rozzano
  - Sandoz Investigational Site, Siena
  - Sandoz Investigational Site, Turin
- Lithuania (2):
  - Sandoz Investigational Site, Kaunas
  - Sandoz Investigational Site, Vilnius
- Malaysia (4):
  - Sandoz Investigational Site, Johor Bahru
  - Sandoz Investigational Site, Kuala Lumpur
  - Sandoz Investigational Site, Pulau Pinang
  - Sandoz Investigational Site, Putrajaya
- Philippines (2):
  - Sandoz Investigational Site, Bacolod
  - Sandoz Investigational Site, Quezon City
- Poland (3):
  - Sandoz Investigational Site, Bydgoszcz
  - Sandoz Investigational Site, Poznan
  - Sandoz Investigational Site, Warsaw
- Portugal (3):
  - Sandoz Investigational Site, Almada
  - Sandoz Investigational Site, Lisbon
  - Sandoz Investigational Site, Porto
- Romania (3):
  - Sandoz Investigational Site, Bucharest
  - Sandoz Investigational Site, Cluj-Napoca
  - Sandoz Investigational Site, Craiova
- South Korea (5):
  - Sandoz Investigational Site, Busan
  - Sandoz Investigational Site, Daegu
  - Sandoz Investigational Site, Daejeon
  - Sandoz Investigational Site, Seoul
  - Sandoz Investigational Site, Suwon
- Spain (13):
  - Sandoz Investigational Site, Barcelona
  - Sandoz Investigational Site, Córdoba
  - Sandoz Investigational Site, Granada
  - Sandoz Investigational Site, Lugo
  - Sandoz Investigational Site, Madrid
  - Sandoz Investigational Site, Marbella
  - Sandoz Investigational Site, Málaga
  - Sandoz Investigational Site, Murcia
  - Sandoz Investigational Site, Oviedo
  - Sandoz Investigational Site, Santa Cruz de Tenerife
  - Sandoz Investigational Site, Santander
  - Sandoz Investigational Site, Santiago de Compostela
  - Sandoz Investigational Site, Valencia
- Taiwan (3):
  - Sandoz Investigational Site, Taichung
  - Sandoz Investigational Site, Tainan
  - Sandoz Investigational Site, Taoyuan

IPD SHARING:
Plan to Share IPD: No